CLINICAL TRIAL: NCT07131176
Title: Assessing the Feasibility of Multimedia Interventions to Reduce Blood Pressure in Marginalized Hypertensive Communities of Karachi, Pakistan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SINA Health Education and Welfare Trust (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 00007
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Cardio Vascular Disease; Educational Intervention; Self Care; Video Streaming
Keywords: high blood pressure; self-care; hypertension; I-changed model; marginalized population; educational intervention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: In the proposed intervention, masking and blinding are essential components to minimize bias and ensure the integrity of the study results. The biostatistician involved in data analysis will be blinded to group assignments, meaning they will not have knowledge of which participants received the video messaging and visual infographics intervention versus those in the control group. This approach prevents any unconscious influence on the statistical analysis, maintaining objectivity in interpreting the outcomes. Additionally, the outcome assessors, who will measure the participants' blood pressure and other health indicators, will also be masked to the group allocations. They will conduct assessments without knowledge of whether the participant is in the intervention or control group, further reducing the risk of bias in the measurement process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Arm: Standardized clinic care with Doctor Advice (No Intervention): In this arm, patient will receive all doctor's consultation and standardized care provided in the clinic setting.
- Intervention :" Educational Intervention through pictorial infographs" (Experimental): Standardized clinic care + pictorial info-graphs distribution at every follow-up visit
  Interventions: Other: Behavior Change through Education intervention
- Intervention : "Education intervention through video of self-care in LCD" (Experimental): Standardized clinic care + hypertension care enhanced Video message in the local language at the waiting area through fastening LCD of the designated cluster.
  Interventions: Other: Behavior Change through Education intervention
- Intervention: Education intervention through video of self-care in LCD + pictorial infograph (Experimental): Standardized clinic care + Hypertension care enhanced pictorial infographic pamphlet distribution at every follow-up visit + hypertension care enhanced Video message at waiting area through fastened LCD of the designated cluster
  Interventions: Other: Behavior Change through Education intervention

INTERVENTIONS:
Other: Behavior Change through Education intervention — The I-Change Model We used behavior alteration theory to identify areas of thinking or conduct that might potentially lead to issues in the process of collecting or consuming medicine. Subsequently, we proceeded to create and improve the substance of the message, and we aligned the messages with a standardized classification of evidence-based strategies for modifying behavior.
  Unclear or confusing information in infographics and television videos was revised, while information that was deemed unhelpful or insignificant by both patients and clinicians was eliminated. Patients' feedback was used to create fresh material for television videos and infographics.
  1. Encourage patients about routine clinic appointments
  2. Provide relevant health-related information.
  3. Help participants plan and organize various treatment adherence behaviors including medication collection and taking, diet, and exercise
  4. Support positive adherence-related behaviors
  Arms: Intervention : "Education intervention through video of self-care in LCD"; Intervention :" Educational Intervention through pictorial infographs"; Intervention: Education intervention through video of self-care in LCD + pictorial infograph

SUMMARY:
This study utilizes the I-Change Model to empower individuals in literacy-limited settings, where the majority of the population is illiterate. By leveraging multimedia tools-such as an educational video and a pictorial infographic-we aim to promote self-care practices among individuals suffering from hypertension. Through these tailored interventions, we seek to enhance awareness, improve hypertension management, and encourage behavioral change, even in low-literacy communities

DETAILED DESCRIPTION:
This study is grounded in the I-Change Model, a behavioral change framework that emphasizes awareness, motivation, and ability as key drivers for adopting healthier lifestyles. Recognizing the barriers posed by low literacy in many underserved communities, particularly in urban slums, we aim to implement context-sensitive interventions that empower individuals with hypertension to take charge of their health. In these settings, traditional written health education materials often fail to reach or resonate with the population due to widespread illiteracy and limited health literacy. To address this gap, our study introduces two key multimedia tools: an educational video, designed with simple language and culturally relevant visuals to demonstrate self-care techniques; and a pictorial infographic that visually conveys essential information about hypertension management, medication adherence, dietary habits, and physical activity. By combining these tools with physician consultations, we hope to strengthen patient understanding, increase engagement with self-care practices, and ultimately improve blood pressure control. This multimedia-based, patient-centered approach offers a scalable and cost-effective strategy for promoting behavioral change in marginalized, low-literacy populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be hypertension patients with an active primary healthcare clinic registration from eight chosen clinics situated in Karachi, Pakistan's slums.
* Anyone between the ages of 21 and 70 who has been diagnosed with hypertension at one of SINA's participating clinics in the last 30 days is eligible to participate.
* Participants will be required to take medicine to control their blood pressure,
* sign an informed consent form,
* attend primary healthcare clinic on a regular basis, and
* have proficiency in five local languages: Urdu, Sindhi, Balochi, Pashto, or Punjabi.

Exclusion Criteria:

* a patient's pregnancy or lactation status, a history of cancer that may necessitate medication changes,
* a blood pressure reading greater than 220/120 mmHg,
* a disability that prevents the patient from reading, writing, communicating, or watching television, and participation in any other study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic and/or Diastolic Blood Pressure | 3, 6, 9 months post intervention
  Change in Systolic and/or Diastolic Blood Pressure from baseline to follow-up

SECONDARY OUTCOMES:
Change in hypertension knowledge score | at 3, 6, 9 months post intervention
  From baseline to post intervention, knowledge about self-care among interventional arms
Adherence to antihypertensive medication | at 3, 6, 9 months post intervention
  The Hill bone-scale, comprising 14 items, assesses medication self-efficacy in managing Hypertension (chronic diseases) and appears suitable for individuals with limited literacy skills
Dietary modifications (e.g., reduced salt intake) | at 3, 6, 9 months post intervention
  Dietary modifications (e.g., reduced salt intake)
Number of clinic visits or follow-up consultations | 3, 6, 9 months post intervention
  Number of clinic visits or follow-up consultations
BMI management in Kg/m2 | 3,6,9 months post intervention
  weight control according to height in kg/m2
Smoking control (number of cigarettes per day) | 3, 6, 9 months post intervention
  Smoking control starting from reduction in number of cigarettes per day to complete cessation
Physical activity | 3, 6, 9 months intervention
  time in minutes which shows physically active in a day (in term of walking, yoga, exercise)

IPD SHARING:
Plan to Share IPD: No
There is confidently matter and Organization will not allow to share